CLINICAL TRIAL: NCT07315607
Title: In Vivo Evaluation of the Accuracy of Immediate Screw-Retained Provisional Crowns Prefabricated Using Digital Planning and Fully Guided Surgery
Brief Title: In Vivo Evaluation of the Accuracy of Immediate Screw-Retained Provisional Crowns Fabricated Using Digital Planning and Guided Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Miguel Gómez Polo, Associate Professor of conservative dentistry and prosthodontics, Universidad Complutense de Madrid
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 25/700-E
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Partial Edentulism; Tooth Loss / Rehabilitation
Keywords: Immediate provisionalization; Screw-retained provisional crown; Guided implant surgery; Digital implant planning
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Intervention Model Description: Participants will undergo a single fully guided implant placement procedure, and outcomes will be evaluated by comparing digitally planned and clinically achieved positions within the same individual.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fully Guided Implant Surgery With Immediate Prefabricated Provisional Crown (Experimental): Participants will undergo a fully guided implant placement procedure with rotational control, followed by the immediate placement of a previously fabricated screw-retained provisional crown designed during the digital planning phase.
  Interventions: Procedure: Fully Guided Implant Placement and Immediate Provisionalization

INTERVENTIONS:
Procedure: Fully Guided Implant Placement and Immediate Provisionalization — Fully guided implant placement using a digitally designed surgical guide with rotational control, followed by immediate placement of a prefabricated screw-retained provisional crown based on the virtual treatment plan.

SUMMARY:
This clinical trial aims to evaluate the in vivo accuracy of a fully digital workflow for the immediate placement of a previously fabricated screw-retained provisional crown using digital planning and guided implant surgery. The study will be conducted in partially edentulous adult patients requiring the replacement of a single tooth with an immediately loaded dental implant.

The main objective of the study is to assess the accuracy (trueness and precision) of the planned digital implant position and provisional restoration by comparing the virtually planned position with the actual clinical outcome after guided surgery. Emphasis will be placed on linear, angular, and rotational deviations at both the implant and provisional restoration levels.

Participants will undergo a fully guided implant placement procedure with rotational control, followed by the immediate placement of a prefabricated screw-retained provisional crown designed during the digital planning phase. Postoperative intraoral scans will be obtained to register the final implant and restoration positions.

The planned and achieved positions will be compared using three-dimensional analysis software to quantify deviations and determine whether the accuracy achieved remains within clinically acceptable limits.

DETAILED DESCRIPTION:
Background Computer-guided implant surgery has consolidated a prosthetically driven approach, in which implant positioning is planned according to the definitive or provisional restoration. The integration of cone-beam computed tomography (CBCT) and intraoral scanning allows for virtual planning of implant position, axis, and prosthetic emergence. However, the accurate transfer of the digital plan to the clinical setting remains subject to cumulative errors throughout the digital and surgical workflow.

Accuracy in guided implant surgery is commonly assessed by comparing the planned and postoperative implant positions using linear and angular deviation metrics. From a clinical perspective, the accuracy at the level of the provisional restoration is of particular relevance, as the restoration must seat passively without requiring significant adjustment. This requirement becomes especially critical when an immediate prefabricated screw-retained provisional crown is placed at the time of surgery, as both positional and rotational accuracy are essential for proper seating.

Recent digital workflows have demonstrated the feasibility of designing and fabricating immediate provisional restorations prior to surgery. The use of guided surgical protocols incorporating rotational control aims to reproduce the planned implant orientation and facilitate the immediate placement of prefabricated restorations. However, the accuracy achievable with such workflows has not been sufficiently quantified in clinical settings.

Justification Despite advances in guided surgery and digital manufacturing, limited clinical evidence exists regarding the accuracy of workflows that combine fully guided implant placement with rotational control and the immediate placement of a prefabricated screw-retained provisional crown. Quantifying plan-to-actual deviations at both the implant and restoration levels is essential to determine the clinical feasibility, predictability, and potential optimization of this protocol.

Study Design This is a prospective, single-arm interventional clinical trial with an intraindividual comparison between the digitally planned implant and provisional restoration positions and the actual clinical outcomes obtained after guided surgery.

Participants The study population will consist of partially edentulous patients aged 18 years or older who require the replacement of a single tooth with an immediately loaded dental implant. All participants must meet the predefined inclusion criteria and none of the exclusion criteria and must provide written informed consent prior to participation.

Intervention All participants will undergo a fully digital workflow including CBCT acquisition, intraoral scanning, virtual implant planning, and the design and fabrication of a surgical guide and a prefabricated screw-retained provisional crown. Implant placement will be performed using a fully guided surgical protocol with rotational control. The provisional restoration will be placed immediately after implant insertion and kept free of occlusal contacts.

Outcome Assessment Postoperative intraoral scans will be obtained with a scan body and with the provisional restoration in place. Three-dimensional analysis software will be used to compare the planned and achieved positions. Linear and angular deviations at the coronal and apical implant levels, as well as deviations of the provisional restoration, will be calculated to assess accuracy in terms of trueness and precision.

Statistical Analysis Descriptive statistics will be used to summarize the deviation measurements. Normality will be assessed, and appropriate parametric or non-parametric tests will be applied to determine whether the observed deviations differ significantly from clinically acceptable thresholds.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older.
2. Partially edentulous patients requiring replacement of a single tooth with an immediately loaded dental implant.
3. Patients classified as ASA I or ASA II according to the American Society of Anesthesiologists physical status classification.
4. Patients with clinical conditions allowing immediate implant placement with a minimum primary stability of ≥25 Ncm.
5. Ability to understand the study procedures and provide written informed consent.
6. Willingness to comply with the study protocol and attend required clinical visits.

Exclusion Criteria:

1. Patients classified as ASA III or ASA IV, or with uncontrolled systemic conditions that may interfere with study participation.
2. Presence of psychiatric or cognitive disorders that may compromise informed consent or protocol compliance.
3. Inability to comply with the visit schedule or required evaluations.
4. Any other condition that, in the investigator's judgment, could compromise patient safety, protocol adherence, or data validity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Implant and Provisional Crown Placement | Immediate postoperative period
  Accuracy will be assessed as the combination of trueness and precision by quantifying plan-to-actual deviations between the digitally planned and clinically achieved implant position and provisional crown position. Linear deviations at the coronal and apical implant levels, angular deviation of the implant axis, and linear and angular deviations of the provisional restoration will be calculated using three-dimensional analysis software.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A Gómez Polo, DDS, PhD, Principal Investigator — Universidad Complutense de Madrid; Juan Ballesteros- Martinez, DDs, MSc, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Complutense University of Madrid, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical and privacy considerations. The data collected include detailed clinical and radiographic information that could potentially allow re-identification of participants, even after de-identification. Data will be used solely for the purposes defined in the approved study protocol.

REFERENCES:
- [Background] Adams CR, Ammoun R, Deeb GR, Bencharit S. Influence of Metal Guide Sleeves on the Accuracy and Precision of Dental Implant Placement Using Guided Implant Surgery: An In Vitro Study. J Prosthodont. 2023 Jan;32(1):62-70. doi: 10.1111/jopr.13503. Epub 2022 Mar 22. PMID 35257456
- [Background] Ballesteros J, Vasquez-Ramos S, Revilla-Leon M, Gomez-Polo M. Immediate placement of a previously manufactured interim screw-retained implant-supported crown by using the implant position determined in the guided implant planning. J Prosthet Dent. 2025 Oct;134(4):908-913. doi: 10.1016/j.prosdent.2025.07.009. Epub 2025 Jul 30. PMID 40744851
- [Background] Yeager B, Cakmak G, Zheng F, Johnston WM, Yilmaz B. Error analysis of stages involved in CBCT-guided implant placement with surgical guides when different printing technologies are used. J Prosthet Dent. 2024 Nov;132(5):995-1004. doi: 10.1016/j.prosdent.2022.11.018. Epub 2023 Jan 21. PMID 36690552
- [Background] Younis H, Lv C, Xu B, Zhou H, Du L, Liao L, Zhao N, Long W, Elayah SA, Chang X, He L. Accuracy of dynamic navigation compared to static surgical guides and the freehand approach in implant placement: a prospective clinical study. Head Face Med. 2024 May 14;20(1):30. doi: 10.1186/s13005-024-00433-1. PMID 38745297
- [Background] Espona J, Roig E, Ali A, Roig M. Immediately loaded interim complete-arch implant-supported fixed dental prostheses fabricated with a completely digital workflow: A clinical technique. J Prosthet Dent. 2020 Oct;124(4):423-427. doi: 10.1016/j.prosdent.2019.08.008. Epub 2019 Dec 18. PMID 31862143
- [Background] Hernandez-Margarit P, Palacios-Banuelos R, Roig M, Altuna P, Blasi A. Digital workflow for designing an interim implant-supported restoration with an optimal emergence profile in an open-source software program. J Prosthet Dent. 2024 Nov;132(5):857-862. doi: 10.1016/j.prosdent.2022.10.013. Epub 2022 Dec 6. PMID 36494239
- [Background] Shah NP, Khanna A, Pai AR, Sheth VH, Raut SR. An evaluation of virtually planned and 3D-printed stereolithographic surgical guides from CBCT and digital scans: An in vitro study. J Prosthet Dent. 2022 Sep;128(3):436-442. doi: 10.1016/j.prosdent.2020.12.035. Epub 2021 Feb 12. PMID 33583616
- [Background] Chen Z, Li J, Ceolin Meneghetti P, Galli M, Mendonca G, Wang HL. Does guided level (fully or partially) influence implant placement accuracy at post-extraction sockets and healed sites? An in vitro study. Clin Oral Investig. 2022 Aug;26(8):5449-5458. doi: 10.1007/s00784-022-04512-y. Epub 2022 May 2. PMID 35499656
- [Background] Werny JG, Frank K, Fan S, Sagheb K, Al-Nawas B, Narh CT, Schiegnitz E. Freehand vs. computer-aided implant surgery: a systematic review and meta-analysis-part 1: accuracy of planned and placed implant position. Int J Implant Dent. 2025 May 2;11(1):35. doi: 10.1186/s40729-025-00622-w. PMID 40314873
- [Background] Putra RH, Yoda N, Astuti ER, Sasaki K. The accuracy of implant placement with computer-guided surgery in partially edentulous patients and possible influencing factors: A systematic review and meta-analysis. J Prosthodont Res. 2022 Jan 11;66(1):29-39. doi: 10.2186/jpr.JPR_D_20_00184. Epub 2021 Jan 26. PMID 33504723
- [Background] Khaohoen A, Powcharoen W, Sornsuwan T, Chaijareenont P, Rungsiyakull C, Rungsiyakull P. Accuracy of implant placement with computer-aided static, dynamic, and robot-assisted surgery: a systematic review and meta-analysis of clinical trials. BMC Oral Health. 2024 Mar 21;24(1):359. doi: 10.1186/s12903-024-04033-y. PMID 38509530
- [Background] Lo Russo L, Ercoli C, Guida L, Merli M, Laino L. Surgical guides for dental implants: Measurement of the accuracy using a freeware metrology software program. J Prosthodont Res. 2023 Apr 12;67(2):300-304. doi: 10.2186/jpr.JPR_D_22_00069. Epub 2022 Aug 11. PMID 35965064
- [Background] Gomez-Polo M, Ballesteros J, Padilla PP, Pulido PP, Revilla-Leon M, Ortega R. Merging intraoral scans and CBCT: a novel technique for improving the accuracy of 3D digital models for implant-supported complete-arch fixed dental prostheses. Int J Comput Dent. 2021 Jun 4;24(2):117-123. PMID 34085497
- [Background] Derksen W, Wismeijer D, Flugge T, Hassan B, Tahmaseb A. The accuracy of computer-guided implant surgery with tooth-supported, digitally designed drill guides based on CBCT and intraoral scanning. A prospective cohort study. Clin Oral Implants Res. 2019 Oct;30(10):1005-1015. doi: 10.1111/clr.13514. Epub 2019 Sep 9. PMID 31330566
- [Background] Kernen F, Kramer J, Wanner L, Wismeijer D, Nelson K, Flugge T. A review of virtual planning software for guided implant surgery - data import and visualization, drill guide design and manufacturing. BMC Oral Health. 2020 Sep 10;20(1):251. doi: 10.1186/s12903-020-01208-1. PMID 32912273
- [Background] Shi Y, Wang J, Ma C, Shen J, Dong X, Lin D. A systematic review of the accuracy of digital surgical guides for dental implantation. Int J Implant Dent. 2023 Oct 25;9(1):38. doi: 10.1186/s40729-023-00507-w. PMID 37875645
- [Background] Bruno V, Badino M, Riccitiello F, Spagnuolo G, Amato M. Computer guided implantology accuracy and complications. Case Rep Dent. 2013;2013:701421. doi: 10.1155/2013/701421. Epub 2013 Sep 3. PMID 24083034
- [Background] Chackartchi T, Romanos GE, Parkanyi L, Schwarz F, Sculean A. Reducing errors in guided implant surgery to optimize treatment outcomes. Periodontol 2000. 2022 Feb;88(1):64-72. doi: 10.1111/prd.12411. PMID 35103317
- [Background] Nulty A. A literature review on prosthetically designed guided implant placement and the factors influencing dental implant success. Br Dent J. 2024 Feb;236(3):169-180. doi: 10.1038/s41415-024-7050-3. Epub 2024 Feb 9. PMID 38332076